CLINICAL TRIAL: NCT05398510
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Intravenous/Subcutaneous Injection of SHR-2010 in Healthy Subjects: a Randomized, Double-blind, Dose-increasing, Placebo-controlled Phase I Clinical Trial
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics Pharmacodynamics of SHR-2010 by Intravenously/Subcutaneously in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-2010-101
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: SHR-2010 injection compared with placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment for intravenously/subcutaneously (Experimental): Treatment for intravenously: 6 dose groups； Treatment for subcutaneously: 3 dose groups.
  Interventions: Drug: SHR-2010 injection
- Placebo for intravenously/subcutaneously (Placebo Comparator): Treatment for intravenously: 6 dose groups； Treatment for subcutaneously: 3 dose groups.
  Interventions: Drug: SHR-2010 injection placebo

INTERVENTIONS:
Drug: SHR-2010 injection — Treatment for intravenously: 6 subjects for SR-2010 injection. Treatment for subcutaneously: 8 subjects for SR-2010 injection.
  Arms: Treatment for intravenously/subcutaneously
Drug: SHR-2010 injection placebo — Treatment for intravenously: 2 subjects for placebo. Treatment for subcutaneously: 2 subjects for placebo.
  Arms: Placebo for intravenously/subcutaneously

SUMMARY:
The study is being conducted to Evaluate the Safety, Tolerability and Pharmacokinetics pharmacodynamics of SHR-2010 by intravenously/subcutaneously in Healthy Subject.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Male or non-pregnant, non-lactating female ages 18 to 55 years old.
3. Weight ≥ 45 kg, and body mass index (BMI) must range from 18 to 28 kg/m2 .
4. Healthy subjects as determined by absence of clinically significant abnormalities on medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory tests performed at screening or baseline period.
5. Subjects must be willing to use a highly effective method of contraception as deemed appropriate by the investigator throughout the study and for at least 3 months after the last study drug administration.

Exclusion Criteria:

1. Evidence or history of serious cardiovascular, hepatic, renal, gastrointestinal, psychiatric, neurological, haematological, or metabolic diseases within 5 years.
2. Subjects with tuberculosis diagnosed by Interferon Gamma Release Assays (IGRA) or chest X-ray.
3. Subjects had any surgery within the past 6 months before screening or planned to undergo surgery during the study period.
4. Estimated Glomerular Filtration Rate（eGFR）<90 mL/min/1.73m2.
5. Positive for hepatitis (including hepatitis B and C), HIV or syphilis at screening.
6. Systolic blood pressure (SBP) > 140 mm Hg or < 90 mm Hg, or diastolic blood pressure (DBP) > 90 mm Hg or < 60 mm Hg and has been considered clinically significant.
7. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or gamma-glutamyl transferase (GGT) ≥2.0 x ULN, or total bilirubin ≥1.5 x ULN.
8. Clinically significant abnormal 12-lead ECG at screening (male with QTcF > 450 ms or female with QTcF > 470 ms).
9. Female subjects who had unprotected sexual behaviour within 14 days before screening.
10. Positive for alcohol breath test at screening or baseline period.
11. Positive urinary drug test at screening or baseline period.
12. Blood collection is difficult or cannot tolerate venipuncture blood collection.
13. Allergic to any ingredient or component in the study drug.
14. Subjects who have taken any prescription drugs, over-the-counter drugs, or Chinese herbal medicine within 14 days prior to using the study drug.
15. Subjects who smoked more than 5 cigarettes daily in the 1 month before screening.
16. History of regular alcohol consumption exceeding 3 units/day for women or 5 units/day for men, more than twice per week (1 unit = 150 ml of beer or 50 ml of wine or 17 ml of alcoholic spirits) within 3 months before screening.
17. Participated in any other clinical trials of any drug or medical device within 3 months before screening.
18. Donated blood or blood products or had substantial loss of blood (more than 400 mL) within 1 month before screening, or received any blood or blood products within 2 months prior to screening.
19. Subjects who received live (attenuated) vaccine within 1 month prior to screening or consider getting a vaccination during the study.
20. The employee of investigator or study centre, with direct involvement in the proposed study.
21. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of subjects with adverse events (AEs) | Baseline up to Day 85
  Incidence of AEs, including any abnormal findings in vital signs, and/or physical examination and/or clinical laboratory assessments and/or 12-lead ECG evaluation and/or IGRA.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: AUC0-t for SHR-2010 | Baseline up to Day 85
  AUC0-t: Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration
Pharmacokinetics (PK) parameter: AUC0-∞ for SHR-2010 | Baseline up to Day 85
  AUC0-∞: Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics (PK) parameter: Cmax for SHR-2010 | Baseline up to Day 85
  Cmax: Maximum plasma concentration
Pharmacokinetics (PK) parameter: Tmax for SHR-2010 | Baseline up to Day 85
  Tmax: Time to reach maximum plasma concentration
Pharmacokinetics (PK) parameter: t1/2 for SHR-2010 | Baseline up to Day 85
  t1/2: Terminal half-life
Pharmacokinetics (PK) parameter: CL of SHR-2010 for administration intravenously | Baseline up to Day 85
  CL: Clearance
Pharmacokinetics (PK) parameter: CL/F of SHR-2010 for administration subcutaneously | Baseline up to Day 85
  CL/F: Apparent clearance
Pharmacokinetics (PK) parameter: V of SHR-2010 for administration intravenously | Baseline up to Day 85
  V: Volume of distribution
Pharmacokinetics (PK) parameter: V/F of SHR-2010 for administration subcutaneously | Baseline up to Day 85
  V/F: Apparent volume of distribution
Pharmacokinetics (PK) parameter: Bioavailability (F) of SHR-2010 | Baseline up to Day 85
  Bioavailability of SHR-2010 for administration subcutaneously.
Pharmacodynamics (PD): C4b level in the serum | Baseline up to Day 85
  C4b level in the serum.
Immunogenicity: Proportion of anti-drug antibodies (ADA) positive subjects | Baseline up to Day 85
  Proportion of anti-drug antibodies (ADA) positive subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin P, Wang C, Hu X, Fang L, Lin H, Sun F, Huang R, Ban R, Feng S, Gao Z, Shen K, Cao Y. Safety, tolerability, pharmacokinetics, and pharmacodynamics of SHR-2010, a novel anti-MASP-2 antibody, in healthy volunteers: a randomized, double-blind, placebo-controlled phase 1 study. Expert Opin Investig Drugs. 2025 Apr;34(4):339-348. doi: 10.1080/13543784.2025.2500291. Epub 2025 May 1. PMID 40297949
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639